CLINICAL TRIAL: NCT06153186
Title: Flunarizine for Treatment Resistant Absence Epilepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The enrollment wasn't as predicted. We didn't have enough numbers to show statistical significance.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mary Connolly, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H19-00185
Record Dates: First submitted 2019-10-29; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Childhood Absence Epilepsy; Juvenile Absence Epilepsy; Juvenile Myoclonic Epilepsy
MeSH Terms: conditions — Epilepsy, Absence; Myoclonic Epilepsy, Juvenile | interventions — Flunarizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Flunarizine (Experimental): Flunarizine 5 mg capsules will be administered once a day at night. If the 5mg/day dose is tolerated by any given participant, the dose will be escalated to 10mg/day taken as two 5mg capsules at night
  Interventions: Drug: Flunarizine Hydrochloride

INTERVENTIONS:
Drug: Flunarizine Hydrochloride — Flunarizine tablet

SUMMARY:
This is an open-label, single-centre study to evaluate the clinical efficacy, safety and tolerability of Flunarizine administered as adjunctive treatment in participants diagnosed with treatment resistant absence epilepsy. The study goal is to see how efficient and safe flunarizine is at decreasing the frequency of absence seizures in children with treatment-resistant refractory epilepsy at doses of 5mg and 10mg once daily.

DETAILED DESCRIPTION:
Flunarizine (flunarizine hydrochloride) is indicated for prophylaxis of migraine (with and without aura) in patients with frequent and severe attacks, who have not responded to other treatment and/or in whom other therapy has resulted in unacceptable side effects. Flunarizine readily crosses the blood brain barrier and its primary mechanism of action is to preferentially block the entry of calcium under pathophysiological conditions preventing cellular calcium overload by reducing excessive transmembrane calcium influx.

Flunarizine has been used successfully for many years in children with migraines and is a firstline, though off-label, treatment for alternating hemiplegia of childhood. It is not labeled for the control of seizures, but has been safely trialed as an anti-seizure medication with promising results.

The primary objective is to assess the efficacy, safety and tolerability of flunarizine compared to a baseline period on absence seizures in patients with treatment refractory epilepsy taking a minimum of one anti-seizure medication (ASM). The primary outcome measure is median percent change in weekly absence seizure frequency in patients treated with flunarizine compared with the baseline period.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 4 to 18 years of age
* Participant has treatment resistant absence seizures. Treatment resistant absence seizures are defined as failure to respond to 2 or more appropriate anti-seizure medications (ASMs). The potential participant must have failed to respond to or tolerate appropriate doses of two of the following: ethosuximide (>/= 20 mg/kg/day), Valproic acid/divalproex sodium (>/= 15 mg/kg/day) or lamotrigine, (>/= 5 mg/kg/day).
* Participant must currently be taking a minimum of one ASM
* Normal development (may have specific learning disabilities and/or attention deficit hyperactivity disorder/attention deficit disorder (ADHD/ADD))
* EEG confirmation of absence seizures and EEG within 2 months of screening visit
* Absence seizures reported at least 10 times per week
* Participants must have no changes in baseline ASMs for 1 month prior to screening period
* Participant or caregiver can maintain a seizure diary
* Participant is able to swallow capsules
* Written informed consent must be provided. Legal guardians of the participants must be able to understand and provide written consent on behalf of the participant, since study participants may be too young to provide informed consent. For participants 7-18 years of age, assent will be required along with written informed consent of the caregiver.
* The participant is willing and able to attend all study visits at British Columbia (BC) Children's Hospital
* Participant has the ability to speak and read in English
* Females of child bearing potential who are sexually active must be willing to use contraceptive methods for the duration of the study and 6 months post last dose of study drug.
* Males who are sexually active with females of child bearing potential must be willing to use contraception for the duration of the study and 3 months post last dose of study drug.

Exclusion Criteria:

* Age < 4 years, > 18 years
* Participant has uncontrolled myoclonic or generalized tonic clonic seizures
* Psychogenic non-epileptic seizures
* Known diagnosis of intellectual disability
* Autism spectrum disorder
* Participant is taking carbamazepine, oxcarbazepine, phenytoin, eslicarbazepine, or vigabatrin
* History of poor compliance with medication
* Inability of parent or caregiver to maintain a seizure diary
* History of depression or psychosis
* Participant has previously taken flunarizine and has had an adverse reaction to treatment
* Participants who are pregnant or breastfeeding,
* Presence of extrapyramidal symptoms
* Participants who have clinically significant hepatic impairment as assessed by the investigator
* Participants with known hypersensitivity to flunarizine or any of its ingredients

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Median Percent Change in Weekly absence seizure frequency | 12 weeks
  Measuring the median percent change in weekly absence seizure frequency in patients treated with flunarizine compared with the baseline period. This will be measured by evaluating patient seizure diaries at baseline and at the end of the treatment period

SECONDARY OUTCOMES:
Evaluating EEG changes in patients with absence epilepsy | 12 weeks
  Median percent change in the number of absence seizures captured on EEG, and bursts of spike/wave lasting 2 or more seconds in patients treated with flunarizine compared with the baseline period

CONTACTS AND LOCATIONS:
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada